CLINICAL TRIAL: NCT03314350
Title: Prevalence of Wound Healing Disturbances in Geriatric Inpatients With Specific Focus on Malnutrition, Other Nutritional Parameters and the Frailty Syndrome (WONDER Study)
Brief Title: Prevalence of Wound Healing Disturbances in Geriatric Inpatients (WONDER Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Kristina Norman, PD Dr. Kristina Norman, Charite University, Berlin, Germany
Other Study IDs: WONDER
Record Dates: First submitted 2017-10-16; First posted 2017-10-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Wound Healing Disorder; Malnutrition
Keywords: Geriatrics; Frailty
MeSH Terms: conditions — Malnutrition; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In geriatric patients, there is a plethora of nutritional and illness-related parameters, resulting in a complex situation which hampers identification of risk factors.In the planned prospective study, the point and period prevalence of wound healing disorders (WHD) is examined at admission and at discharge in a cohort of 517 male and female geriatric patients. As the investigators are also interested to study the occurrence of WHD in patients with malnutrition (and other geriatric phenomena) compared to the prevalence of WHD in patients with a good nutritional Status.

DETAILED DESCRIPTION:
The investigators will determine the prevalence of impaired wound healing upon admission to the hospital as well as the incidence of new wound healing disorders during hospital stay with specific focus on malnutrition and other important nutritional parameters in geriatric patients. Therefore the investigators intend to study consecutively admitted patients both at admission and at discharge and monitor them during hospital stay.

The investigators will investigate the associations between the individual nutritional status and body composition parameters (such as sarcopenia) and WHD in geriatric patients, taking both medical variables and the frailty syndrome into account.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Informed written consent
* Normal cognitive status according to Mini-Mental State Examination (MMSE ≥ 24 points)
* Life expectancy of > 3 months according to treating doctor
* Proficient in German

Exclusion Criteria:

* Lack or incapacity of informed consent
* MMSE < 24
* Life expectancy < 3 months according to assessment by the attending physician
* Short term patients (< 3 days of hospital stay)
* Lack of German language

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Geriatric patients will be recruted upon admission to the hospital.
Sampling Method: Probability Sample
Enrollment: 517 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of wound healing disturbances | Baseline
  Number of wound healing disturbances upon admission to the hospital in General

SECONDARY OUTCOMES:
Nutritional Parameter | Baseline and up to 3 weeks
  Mini Nutritional Assessment - Short Form (questionnaire)
Functional Parameter | Baseline and up to 3 weeks
  Timed Up & Go Test
Functional Parameter | Baseline and up to 3 weeks
  4m-walk Test to measure gait speed
Functional Parameter | Baseline and up to 3 weeks
  Lung Test to measure respiratory force
Strength Parameter | Baseline and up to 3 weeks
  Hand grip strength
Strength Parameter | Baseline and up to 3 weeks
  Knee extension strength
Frailty | Baseline and up to 3 weeks
  Frailty Status according to Fried criteria
Index of quality of life | Baseline and up to 3 weeks, after 3 months and after 6 months
  EQ-5D-5L (questionnaire) to measure quality of life
Body composition | Baseline and up to 3 weeks
  Bioelectric impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Norman, PD Dr., Principal Investigator — Charite Research Group on Geriatrics
Locations (1):
- Charite University Medicine, Research Group on Geriatrics, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shahin ES, Meijers JM, Schols JM, Tannen A, Halfens RJ, Dassen T. The relationship between malnutrition parameters and pressure ulcers in hospitals and nursing homes. Nutrition. 2010 Sep;26(9):886-9. doi: 10.1016/j.nut.2010.01.016. Epub 2010 May 4. PMID 20444575